CLINICAL TRIAL: NCT00904813
Title: A Prospective Randomized Trial on Different Preoperative Radiotherapy Regimens in Rectal Cancer, Stockholm III.
Brief Title: The Stockholm III Trial on Different Preoperative Radiotherapy Regimens in Rectal Cancer
Acronym: Stockholm III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Swedish Cancer Society (Other); The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Anna Martling, Professor, Senior Consultant Surgeon, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 98/240
Record Dates: First submitted 2009-05-19; First posted 2009-05-20 (Estimated); Results first posted 2021-04-06 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-04

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Preoperative radiotherapy; Timing of Surgery; Prognosis
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1. Short-course RT (5x5 Gy) + surgery within 1 week (SRT) (Active Comparator): RT=Preoperative radiotherapy Gy=Gray
  Interventions: Radiation: Short-course RT
- 2. Short-course RT (5x5 Gy) + surgery after 4-8 weeks (SRT-delay) (Active Comparator): RT=Preoperative radiotherapy Gy= Gray
  Interventions: Radiation: Short-course RT
- 3. Long-course RT (25x2 Gy) + surgery after 4-8 weeks (LRT-delay) (Active Comparator): RT= Preoperative radiotherapy Gy= Gray
  Interventions: Radiation: Long-course RT

INTERVENTIONS:
Radiation: Short-course RT — Preoperative radiotherapy (RT) given 5 times 5 Gray during five consecutive days, preferably Monday - Friday, with a four-field box technique, including the primary tumour and the primary and secondary lymph nodes in the pelvis.
  Arms: 1. Short-course RT (5x5 Gy) + surgery within 1 week (SRT); 2. Short-course RT (5x5 Gy) + surgery after 4-8 weeks (SRT-delay)
Radiation: Long-course RT — Preoperative radiotherapy (RT) given 2 Gy in 25 fractions during 5 weeks, total dose 50 Gy with a four-field box technique, including the primary tumour and the primary and secondary lymph nodes in the pelvis.
  Arms: 3. Long-course RT (25x2 Gy) + surgery after 4-8 weeks (LRT-delay)

SUMMARY:
Preoperative radiotherapy (RT) is recommended to many patients with localised rectal cancer, not previously treated with pelvic RT. However, the optimum fractionation, the timing of surgery and the best use of concomitant chemotherapy remains controversial. There are theoretical reasons to believe that radiotherapy given in larger fractions during a shorter period of time might result in more late side effects than giving a conventional, more protracted RT in patients with rectal cancer. In addition, the optimum timing of surgery after RT, with respect to postoperative morbidity, mortality and potential downsizing of the tumour is not known.

To address these questions, a prospective randomized multicenter trial was initiated, the Stockholm III trial, in which patients with primarily resectable rectal cancer were randomized to short-course preoperative RT (5x5 Gy) followed by surgery within one week or after 4-8 weeks or long-course preoperative RT(25x2 Gy) followed by surgery after 4-8 weeks.

DETAILED DESCRIPTION:
840 participants (men and women) with a biopsy verified adenocarcinoma of the rectum scheduled for an open abdominal procedure were enrolled at 18 Swedish Hospitals during 1998-2013.

In the initial protocol patients were randomly assigned (1:1:1) between three different RT courses; 5x5 Gy with surgery within 1 week (SRT), 5x5 Gy with surgery after 4-8 weeks (SRT-delay) or 25x2 Gy during 5 weeks without concomitant chemotherapy and surgery after 4-8weeks (LRT-delay). After a protocol amendment on May 21, 1999, participating hospitals could choose to randomise patients to just the short-course radiotherapy arms (1:1) or to all three arms.

Randomisation was done by telephone by the Regional Cancer Centre in Stockholm, Sweden, after assessing inclusion and exclusion criteria. Computer generated randomisation lists were constructed by use of permuted block technique (block size of six for the three- arm randomisation, block size of four for the two-arm randomisation) and stratified by participating center. Investigators and patients were not masked to treatment.

Follow-up was recommended at 3-, 6- and 12 months after surgery, and yearly thereafter. Although follow-up according to national guidelines with a minimum follow-up at 1 and 3 years was allowed. Patient data was also collected from the Swedish ColoRectal Cancer Register (SCRCR) and medical records.

Primary outcome:

1. Time to local recurrence.

Secondary outcomes:

1. Recurrence-free survival
2. Frequency of postoperative complications
3. Frequency of tumour regression

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed clinically resectable rectal adenocarcinoma within 15 cm from the anal verge
* Planned for bowel resection with an abdominal procedure.
* Informed consent.

Exclusion Criteria:

* Distant metastases
* Locally advanced unresectable tumors
* Planned for local excision
* Previous radiotherapy to the abdominal or pelvic region
* Severe ischemic heart disease or symptoms of severe arteriosclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 1998-11; Primary Completion 2015-02 (Actual); Study Completion 2018-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Martling, Professor, Principal Investigator — Karolinska Institutet
Locations (18):
- Sweden (18):
  - Mora Hospital, Mora, Dalarna County
  - Danderyds Hospital, Danderyd, Stockholm County
  - Norrtälje Hospital, Norrtälje, Stockholm County
  - Södertälje Hospital, Södertälje, Stockholm County
  - Eskilstuna Hospital, Eskilstuna
  - Falun Hospital, Falun
  - Gävle Sjukhus, Gävle
  - Helsingborg Hospital, Helsingborg
  - Linköping University Hospital, Linköping
  - MAS University Hospital, Malmo
  - Vrinnevi Hospital, Norrköping
  - Karolinska University Hospital, Stockholm
  - Ersta Hospital, Stockholm
  - South Hospital, Stockholm
  - St Görans Hospital, Stockholm
  - Norrlands Universitetssjukhus, Umeå
  - Uppsala University Hospital, Uppsala
  - Visby Hospital, Visby

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pettersson D, Lorinc E, Holm T, Iversen H, Cedermark B, Glimelius B, Martling A. Tumour regression in the randomized Stockholm III Trial of radiotherapy regimens for rectal cancer. Br J Surg. 2015 Jul;102(8):972-8; discussion 978. doi: 10.1002/bjs.9811. PMID 26095256
- [Background] Pettersson D, Cedermark B, Holm T, Radu C, Pahlman L, Glimelius B, Martling A. Interim analysis of the Stockholm III trial of preoperative radiotherapy regimens for rectal cancer. Br J Surg. 2010 Apr;97(4):580-7. doi: 10.1002/bjs.6914. PMID 20155787
- [Background] Pettersson D, Glimelius B, Iversen H, Johansson H, Holm T, Martling A. Impaired postoperative leucocyte counts after preoperative radiotherapy for rectal cancer in the Stockholm III Trial. Br J Surg. 2013 Jun;100(7):969-75. doi: 10.1002/bjs.9117. Epub 2013 Apr 2. PMID 23553796
- [Result] Erlandsson J, Holm T, Pettersson D, Berglund A, Cedermark B, Radu C, Johansson H, Machado M, Hjern F, Hallbook O, Syk I, Glimelius B, Martling A. Optimal fractionation of preoperative radiotherapy and timing to surgery for rectal cancer (Stockholm III): a multicentre, randomised, non-blinded, phase 3, non-inferiority trial. Lancet Oncol. 2017 Mar;18(3):336-346. doi: 10.1016/S1470-2045(17)30086-4. Epub 2017 Feb 10. PMID 28190762
- [Result] Erlandsson J, Lorinc E, Ahlberg M, Pettersson D, Holm T, Glimelius B, Martling A. Tumour regression after radiotherapy for rectal cancer - Results from the randomised Stockholm III trial. Radiother Oncol. 2019 Jun;135:178-186. doi: 10.1016/j.radonc.2019.03.016. Epub 2019 Apr 1. PMID 31015165
- [Result] Erlandsson J, Pettersson D, Glimelius B, Holm T, Martling A. Postoperative complications in relation to overall treatment time in patients with rectal cancer receiving neoadjuvant radiotherapy. Br J Surg. 2019 Aug;106(9):1248-1256. doi: 10.1002/bjs.11200. Epub 2019 Jun 14. PMID 31197822

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 18 hospitals in Sweden between 1998-2013 and initially randomly assigned (1:1:1) to three different arms; Short-course radiotherapy with surgery within 1 week (SRT) or after 4-8 weeks (SRT-delay), or Long-course radiotherapy with surgery after 4-8 weeks (LRT-delay). After a protocol amendment in 1999 hospitals could choose to randomise patients to all three arms or only short-course treatment arms (SRT or SRT-delay, 1:1). Patients could only be randomised to one arm.
Pre-assignment Details: Of 8122 eligible patients, 385 were assigned to the three-armed randomisation and 455 to the two-armed randomisation, resulting in 840 participants included in the study.
Groups:
- Three-arm Randomisation: SRT: Participants included in the three-armed randomisation and allocated to short-course preoperative radiotherapy (5x5 Gy) and surgery within 1 week.
- Three-arm Randomisation: SRT-delay: Participants included in the three-armed randomisation and allocated to short-course preoperative radiotherapy (5x5 Gy) and surgery after 4-8 weeks.
- Three-arm Randomisation: LRT-delay: Participants included in the three-armed randomisation and allocated to long-course preoperative radiotherapy (25x5 Gy) and surgery after 4-8 weeks.
- Two-arm Randomisation: SRT: Participants included in the two-armed randomisation and allocated to short-course preoperative radiotherapy (5x5 Gy) and surgery within 1 week.
- Two-arm Randomisation: SRT-delay: Participants included in the two-armed randomisation and allocated to short-course preoperative radiotherapy (5x5 Gy) and surgery after 4-8 weeks.
Period: Overall Study
Arm/Group | Three-arm Randomisation: SRT | Three-arm Randomisation: SRT-delay | Three-arm Randomisation: LRT-delay | Two-arm Randomisation: SRT | Two-arm Randomisation: SRT-delay
Started | 129 | 128 | 128 | 228 | 227
Completed | 129 | 128 | 128 | 228 | 227
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Three-arm Randomisation: SRT | Three-arm Randomisation: SRT-delay | Three-arm Randomisation: LRT-delay | Two-arm Randomisation: SRT | Two-arm Randomisation: SRT-delay | Total
Number analyzed (Participants) | 129 | 128 | 128 | 228 | 227 | 840
Age, Continuous [Median (Full Range); unit: years] | 67 [62 to 74] | 67 [62 to 75] | 66 [61 to 73] | 67 [61 to 74] | 67 [61 to 74] | 67 [61 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 49 | 55 | 91 | 93 | 336
  Male | 81 | 79 | 73 | 137 | 134 | 504
Tumour height from anal verge [Count of Participants; unit: Participants]
  0-5 centimeter | 50 | 57 | 31 | 78 | 68 | 284
  6-10 centimeter | 49 | 49 | 60 | 91 | 95 | 344
  11-15 centimeter | 30 | 21 | 35 | 58 | 63 | 207
  Missing | 0 | 1 | 2 | 1 | 1 | 5
Type of Surgery [Count of Participants; unit: Participants]
  Anterior Resection | 79 | 68 | 93 | 139 | 136 | 515
  Abdominal perineal excision | 47 | 53 | 24 | 75 | 79 | 278
  Hartmann's | 3 | 6 | 8 | 14 | 12 | 43
  Local excision | 0 | 1 | 0 | 0 | 0 | 1
  No resection | 0 | 0 | 3 | 0 | 0 | 3
ypStage [Count of Participants; unit: Participants] — Pathological tumour stage after neoadjuvant treatment calculated according to the AJCC 8th edition. Stages ranging from I to IV with higher number indicating more advanced cancer. Stage x = Unknown stage.
  Participants
    I | 38 | 55 | 37 | 58 | 83 | 271
    II | 43 | 31 | 46 | 75 | 55 | 250
    III | 48 | 31 | 37 | 86 | 76 | 278
    IV | 0 | 7 | 5 | 7 | 6 | 25
    Stage x | 0 | 3 | 1 | 1 | 6 | 11
    Missing | 0 | 1 | 2 | 1 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Time to Local Recurrence.
Description: Local recurrence was defined as tumour growth below the level of the sacral promontory, related to the previous rectal cancer, and diagnosed radiographically with MRI, CT, or both, or clinically (preferably with histological confirmation). A diagnosis of local recurrence was confirmed and reported by the patient-responsible physician to the Swedish ColoRectal Cancer Registry (SCRCR), a nationwide validated national registry. Local recurrence was measured both as first and any event occurring during follow-up (censoring date March 30 2015), when all patients had been followed for at least 2 years.
Time Frame: From date of randomisation until date of local recurrence or date of death from any cause, whichever came first, assessed up to end of follow-up.
Population: Participants were analysed according to intention to treat.
Measure: Median (Full Range); unit: months
Groups:
- Pooled Short-course RT: SRT: Participants assigned to short-course preoperative radiotherapy (5x5 Gy) and surgery within 1 week pooled from the three-armed and two-armed randomisation.
- Pooled Short-course RT: SRT-delay: Participants assigned to short-course preoperative radiotherapy (5x5 Gy) and surgery after 4-8 weeks pooled from the three-armed and two-armed randomisation.
Arm/Group | Three-arm Randomisation: SRT | Three-arm Randomisation: SRT-delay | Three-arm Randomisation: LRT-delay | Two-arm Randomisation: SRT | Two-arm Randomisation: SRT-delay | Pooled Short-course RT: SRT | Pooled Short-course RT: SRT-delay
Number analyzed (Participants) | 129 | 128 | 128 | 228 | 227 | 357 | 355
months | 28.3 [20.7 to 62.2] | 22.1 [15.5 to 34.3] | 33.3 [17.8 to 114.3] | 35.1 [18.2 to 59.9] | 17.2 [8.5 to 39.5] | 33.4 [18.2 to 62.2] | 19.3 [8.5 to 39.5]
Statistical Analysis 1: Comparison: Three-arm Randomisation: SRT vs Three-arm Randomisation: SRT-delay vs Three-arm Randomisation: LRT-delay; The effect of treatment regimen on local recurrence as first event in the three-armed group comparison (n = 385) was estimated with proportional hazards regression, stratified by participating centre; Test type: Non-Inferiority — In the initial protocol treatment groups were deemed non-inferior if the upper limit of a two-sided 90% CI for the hazard ratio did not exceed 1.7. With a cumulative incidence of local recurrence at 15%, a sample size of 840 participants were determined to provide a power of 80%. However, due to lower recurrence rate, the trial was re-powered in the amendment 1999 to deem non-inferiority at an HR not exceeding 2.5 or 3.6 depending on the frequency of local recurrence; p = 0.52, Log Rank — The threshold for statistical significance was p=0.05; An overall p-value was calculated; Hazard Ratio (HR) = 0.38, 90% CI 2-sided [0.06 to 2.56] — SRT was used as reference group. Estimation described above is for SRT-delay. For LRT-delay HR (90% CI) was 1.22 with lower limit: 0.33, and upper limit: 3.45
Statistical Analysis 2: Comparison: Three-arm Randomisation: SRT vs Three-arm Randomisation: SRT-delay vs Three-arm Randomisation: LRT-delay; The effect of treatment regimen on recurrence-free survival in the three armed randomisation comparison (n = 385) was estimated with proportional hazards regression, stratified by participating centre; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.92, Log Rank — The threshold for statistical significance was p=0.05; An overall p-value was calculated; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.64 to 1.35] — SRT was used as reference group (1.00). Estimation described above is for SRT-delay. For LRT-delay HR (95% CI) was 0.99 with lower limit: 0.68, and upper limit: 1.42
Statistical Analysis 3: Comparison: Pooled Short-course RT: SRT vs Pooled Short-course RT: SRT-delay; The effect of treatment regimen on local recurrence as first event in the pooled short-course RT comparison (n = 712) was estimated with proportional hazards regression, stratified by participating centre; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.59, Log Rank — The threshold for statistical significance was p=0.05; Hazard Ratio (HR) = 0.91, 90% CI 2-sided [0.36 to 2.27] — SRT was used as reference group (1.00). Estimation described above is for SRT-delay
Statistical Analysis 4: Comparison: Pooled Short-course RT: SRT vs Pooled Short-course RT: SRT-delay; The effect of treatment regimen on recurrence-free survival in the pooled short-course RT comparison (n = 712) was estimated with proportional hazards regression, stratified by participating centre; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.39, Log Rank — The threshold for statistical significance was p=0.05; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.69 to 1.18] — SRT was used as reference group. Estimation described above is for SRT-delay

2. Secondary Outcome: Number of Participants With Postoperative Complications in Relation to Preoperative Radiotherapy Regimen and Overall Treatment Time.
Description: Postoperative complications was defined as any cardiovascular event, infectious, neurological or surgical complications occurring within 30 days after surgery, or during the same hospital admission, validated from medial records. Overall postoperative complication was defined as having at least one postoperative complication. Participants were grouped based on type of preoperative radiotherapy (RT) regimen (eg short- or long course) and overall treatment time (OTT), defined as time between start of RT and surgery. Participants receiving short-course RT were categorised into four different groups; Group A: OTT 7 days, Group B: OTT 8-13 days, Group C: OTT 5-7 weeks, Group D: OTT 8-13 weeks. Participants receiving long-course RT were categorised into two different groups; Group E: OTT 9-11 weeks, Groups F: OTT 12-14 weeks.
Time Frame: From surgery until 30 days postoperatively.
Population: Participants were analysed as treated and grouped based on type of preoperative radiotherapy (RT) and overall treatment time (OTT).
Measure: Count of Participants; unit: Participants
Groups:
- Group A: Short-course RT and OTT 7 Days: Participants treated with short-course preoperative radiotherapy (5x5 Gy) with overall treatment time of 7 days.
- Group B: Short-course RT and OTT 8-13 Days: Participants treated with short-course preoperative radiotherapy (5x5 Gy) with overall treatment time of 8-13 days.
- Group C: Short-course RT and OTT 5-7 Weeks: Participants treated with short-course preoperative radiotherapy (5x5 Gy) with overall treatment time of 5-7 weeks.
- Group D: Short-course RT and OTT 8-13 Weeks: Participants treated with short-course preoperative radiotherapy (5x5 Gy) with overall treatment time of 8-13 weeks.
- Group E: Long-course RT and OTT 9-11 Weeks: Participants treated with long-course preoperative radiotherapy (25x2 Gy) with overall treatment time 9 -11 weeks.
- Group F: Long-course RT and OTT 12-14 Weeks: Participants treated with long-course preoperative radiotherapy (25x2 Gy) with overall treatment time 12 - 14 weeks.
Arm/Group | Group A: Short-course RT and OTT 7 Days | Group B: Short-course RT and OTT 8-13 Days | Group C: Short-course RT and OTT 5-7 Weeks | Group D: Short-course RT and OTT 8-13 Weeks | Group E: Long-course RT and OTT 9-11 Weeks | Group F: Long-course RT and OTT 12-14 Weeks
Number analyzed (Participants) | 100 | 247 | 192 | 160 | 52 | 59
Participants
  Overall postoperative complications | 45 | 138 | 82 | 63 | 16 | 28
  No postoperative complication | 55 | 109 | 110 | 97 | 36 | 31
Statistical Analysis 1: Comparison: Group A: Short-course RT and OTT 7 Days vs Group B: Short-course RT and OTT 8-13 Days; The association between postoperative complications and short-course RT by overall treatment time was assessed using logistic regression analysis; Test type: Superiority; p = 0.289, Regression, Logistic — The threshold of statistical significance was p=0.05; Model was adjusted for sex, age over 75 years, type of surgery and ASA fitness grade; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.40 to 1.32] — Group B was used as the reference group
Statistical Analysis 2: Comparison: Group B: Short-course RT and OTT 8-13 Days vs Group C: Short-course RT and OTT 5-7 Weeks; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.009, Regression, Logistic — The threshold for statistical significance was p=0.05; Model was adjusted for sex, age over 75 years, type of surgery and ASA fitness grade; Odds Ratio (OR) = 0.5, 95% CI 2-sided [0.30 to 0.84] — Group B was used as the reference group
Statistical Analysis 3: Comparison: Group B: Short-course RT and OTT 8-13 Days vs Group D: Short-course RT and OTT 8-13 Weeks; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Regression, Logistic — The threshold for statistical significance was p-value=0.05; Model was adjusted for sex, age over 75 years, type of surgery and ASA fitness grade; Odds Ratio (OR) = 0.39, 95% CI 2-sided [0.23 to 0.65] — Group B was used as the reference group
Statistical Analysis 4: Comparison: Group E: Long-course RT and OTT 9-11 Weeks vs Group F: Long-course RT and OTT 12-14 Weeks; The association between postoperative complications and long-course RT by overall treatment time was assessed using logistic regression analysis; Test type: Superiority; p = 0.521, Regression, Logistic — The threshold for statistical significance was p-value = 0.05; Model was adjusted for sex, age over 75 years, type of surgery and ASA fitness grade; Odds Ratio (OR) = 1.58, 95% CI 2-sided [0.39 to 6.37] — Group E was used as the reference group

3. Secondary Outcome: Tumour Regression Based on the Dworak Grading Scoring System
Description: Tumour regression (TRG) was assessed using the Dworak grading scoring system, ranging from scores 0 to 4 with higher scores indicating better tumour regression. Definition of scores; 0 = no regression, 1 = dominant tumour mass with obvious fibrosis and/or vasculopathy, 2 = dominantly fibrotic changes with few tumour cells or groups (easy to find), 3 = very few (difficult to find microscopically) tumour cells in fibrotic tissue with or without mucous substance, 4 = no tumour cells, only fibrotic mass (total regression or complete response). All available microscopy slides were assessed by one pathologist, blinded to treatment.
Time Frame: At the time of surgery.
Population: Participants grouped based on allocated treatment and analysed as-treated. Only participants with available microscopy slides were included in the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Short-course RT: SRT: Participants treated with short-course preoperative radiotherapy (5x5 Gy) and surgery within 1 week.
- Short-course RT: SRT-delay: Participants treated with short-course preoperative radiotherapy (5x5 Gy) and surgery after 4-8 weeks.
- Long-course RT: LRT-delay: Participants treated with long-course preoperative radiotherapy (25x5 Gy) and surgery after 4-8 weeks.
Arm/Group | Short-course RT: SRT | Short-course RT: SRT-delay | Long-course RT: LRT-delay
Number analyzed (Participants) | 318 | 285 | 94
Participants
  TRG 0 | 29 | 20 | 4
  TRG 1 | 233 | 124 | 42
  TRG 2 | 50 | 92 | 37
  TRG 3 | 2 | 16 | 7
  TRG 4 | 4 | 29 | 3
  Not assessable | 0 | 4 | 1
Statistical Analysis 1: Comparison: Short-course RT: SRT vs Short-course RT: SRT-delay vs Long-course RT: LRT-delay; The association between pathological complete response (pCR), eg no signs of viable tumour or metastatic nodes (T0N0) and overall survival (OS) was assessed using Cox-regression model; Test type: Superiority; p = 0.046, Regression, Cox — The threshold for statistical significance was p=0.05; Model adjusted for age, sex and type of surgery; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.26 to 0.99] — No pCR was used as reference group

ADVERSE EVENTS:
Description: Serious adverse events: Acute radiation-induced toxicity was not assessed in such manner that specific terms can be separated.
Groups:
- Pooled Short-course RT: SRT: Participants assigned to short-course preoperative radiotherapy (5x5 Gy) and surgery within 1 week pooled from both three-armed and two-armed randomisation.
- Pooled Short-course RT: SRT-delay: Participants assigned to short-course preoperative radiotherapy (5x5 Gy) and surgery after 4-8 weeks pooled from both three-armed and two-armed randomisation.
Arm/Group | Three-arm Randomisation: SRT | Three-arm Randomisation: SRT-delay | Three-arm Randomisation: LRT-delay | Pooled Short-course RT: SRT | Pooled Short-course RT: SRT-delay
All-Cause Mortality (participants affected / at risk) | 51/129 | 43/128 | 49/128 | 110/357 | 108/355
Serious Adverse Events (participants affected / at risk) | 0/129 | 7/128 | 6/128 | 1/357 | 23/355
Other Adverse Events (participants affected / at risk) | 65/129 | 48/128 | 50/128 | 188/357 | 144/355
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Three-arm Randomisation: SRT (N=129) | Three-arm Randomisation: SRT-delay (N=128) | Three-arm Randomisation: LRT-delay (N=128) | Pooled Short-course RT: SRT (N=357) | Pooled Short-course RT: SRT-delay (N=355)
Acute radiation-induced toxicity (Gastrointestinal disorders) | 0 | 7 | 6 | 1 | 23 — Defined as unplanned patient admission to hospital with symptoms of radiation side-effects, corresponding to the Radiotherapy Oncology Group (RTOG) scales 3-4 occurring between radiotherapy initiation and the date of surgery.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Three-arm Randomisation: SRT (N=129) | Three-arm Randomisation: SRT-delay (N=128) | Three-arm Randomisation: LRT-delay (N=128) | Pooled Short-course RT: SRT (N=357) | Pooled Short-course RT: SRT-delay (N=355)
Reoperation (Surgical and medical procedures) | 11 | 7 | 7 | 43 | 37 — Defined as a surgical intervention requiring anaesthesia due to a postoperative complication.
Any postoperative complication (Surgical and medical procedures) | 65 | 48 | 50 | 188 | 144 — Defined as any cardiovascular, infectious, neurological or surgical complication noted within 30 days after surgery.
Any surgical complication (Surgical and medical procedures) | 40 | 33 | 30 | 128 | 100 — Defined as any surgical site infection, deep infection, anastomotic leak, postoperative bleeding, stoma related complications, wound dehiscence, or other surgical complication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes